CLINICAL TRIAL: NCT06613334
Title: Automatic Measurement of Antipsychotic Medication Adherence in Schizophrenia Through Speech (OBSERVSPEECH)
Brief Title: Voice-Based Biomarkers: a Novel Approach to Monitoring and Predicting Schizophrenia Relapses
Acronym: OBSERVSPEECH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D23-P038
Record Dates: First submitted 2024-09-10; First posted 2024-09-25 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: Patients with schizophrenia are assigned prospectively to the following experimental interventions: blood tests to measure antipsychotics concentration and the administration of questionnaires/voice tests on the CALLYOPE application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Schizophrenic patients treated with a primary treatment (Experimental): Study's interventions:
  * 4 blood tests (inclusion visit, at follow-up visits at 2 and 4 months after inclusion, at the end-of-study visit at 6 months after inclusion) to measure the blood concentration of antipsychotic treatment (risperidone or paliperidone)
  * completion of self-questionnaires and voice interviews of the application developed by CALLYOPE
  Interventions: Biological: Blood test: measurement of plasma antipsychotic concentration; Other: Voice interviews and questionnaires carried out via the CALLYOPE application

INTERVENTIONS:
Biological: Blood test: measurement of plasma antipsychotic concentration — Four blood tests are prospectively realized per patient during the study to measure the plasma concentration of antipsychotics (primary treatment: risperidone/paliperidone, olanzapine or aripiprazole). These blood samples are taken at the inclusion visit, at the follow-up visits 2 and 4 months after the inclusion visit, then at the end-of-study visit 6 months after the inclusion visit.
Other: Voice interviews and questionnaires carried out via the CALLYOPE application — Voice interviews carried out via the Callyope application: they consist of a series of tests, divided into two parts: Structured tasks (same content for each participant) and Semi-structured tasks (content varies for each participant).
  The simultaneous analysis of several speech tasks allows us to break down the different stages of speech production and the important factors that influence its achievement.
  In addition, patients will complete self-questionnaires via the application. Finally, lifestyle habits (sleep duration and number of steps) will be recorded via the application.
  These different tests will be carried out on the application at the inclusion visit (M0), then every month (M1, M2, M3, M4, M5) until the end of study visit (M6).

SUMMARY:
Schizophrenia is a serious psychiatric illness affecting approximately 25 million people worldwide. Patients with schizophrenia experience hallucinations, auditory illusions, disordered thinking, movement disorders, cognitive impairment and social isolation. Treatments with antipsychotics have proven effective in improving their living conditions, but poor compliance results in relapses and rehospitalizations for the majority of patients, which often results in a worsening of residual symptoms. The prevention of these relapses is a major issue in the care of these patients and frequent monitoring is necessary. The use of a simple, rapid and inexpensive tool to monitor symptoms and treatment effect in schizophrenia could improve the effectiveness of the treatment of these patients and prevent relapses. Speech is a good candidate as a biomarker in the monitoring of patients with schizophrenia. Schizophrenia is accompanied by speech disorders including poor speech, variations in tone or intensity or even difficulties in organizing speech.

DETAILED DESCRIPTION:
Schizophrenia is a highly complex disease of unknown origin. It is characterized by a heterogeneous etiology and variable clinical manifestations. Numerous studies have investigated genetic, biochemical or neurodevelopmental factors of the pathology, without providing a definitive answer. The environmental factor is also analyzed, especially urban density and pollution. Finally, the immune pathway, in particular neuroinflammation, has been studied. Certain parasites, such as Toxoplasma, may be involved in the development of schizophrenia in combination with genetic factors. All these studies tend to show that the parasite/gene/environment association would influence the development of schizophrenia, but the origins remain unclear and a more complete knowledge of the pathophysiology is needed to improve diagnosis and patient management through new therapeutic targets.

More than 80% of patients with schizophrenia have language abnormalities. These abnormalities are manifested in syntax, semantics and phonology. The most common include monotonous intonation, poverty of speech, increased pauses, lack of spontaneity, and disruption of speech coherence. As speech is an important factor in social interaction, patients have great difficulty in maintaining their social relationships.

A major problem in schizophrenia is the discontinuation or misuse of antipsychotic treatment, which leads to relapse and additional hospital costs. According to a 2013 study, 50% of patients discontinue treatment after six months, often leading to decompensations.To avoid relapses, clinicans can either administer hetero-questionnaire to monitor the patients' symptoms or monitor treatment adherence.

To monitor symptoms, clinicians have at their disposal various standardized questionnaires such as the PAANS. However, those tests are time-intensive.

To monitor treatment adherence, clinicians can use blood drug concentrations as an evidence of compliance, although this method is invasive, and requires costly administration coordination between healthcare profesionnals and patients. There are also several standardized tests to monitor adherence, such as the clinician-administered BARS questionnaire and the self-administered BEMIB. These measures have often been criticized due to factors such as recall bias and poor self-perception, which limit the accuracy of patient reports and overestimate adherence.

It is therefore essential to develop new tools to objectively measure evolution of symptoms and treatment effects to detect onset of relapses, without increasing the burden on patients' daily lives.

Speech voice markers stand out because they have characteristics that make it easy to use in clinical practice and can be easily integrated into patients' daily lives. Advances in signal processing and machine learning algorithms now make it possible to measure the different components of speech: phonatory skills, articulation, the different linguistic levels (semantics, syntax, morphology, pragmatics) as well as the specific disfluencies of spontaneous speech.

These different speech markers have been validated in different neurological and psychiatric pathologies: in particular, Parkinson's disease, Huntington's disease, depression, suicidal risk, and schizophrenia. These markers of speech in psychiatry are now generalizing across languages and are also being taken into patients' homes to measure changes in patient states.

Distinctive voice characteristics have been a feature of schizophrenia since it was first defined. They are often associated with negative symptoms, such as the inability to show emotion, and with observed social impairments. It has been quantitatively observed that people with schizophrenia have poorer speech, more pauses, distinctive tones, and differences in voice intensity.

Studies have shown antipsychotics also affect language, since patients are dopamine-deficient, and blockade of these receptors by antipsychotics would exacerbate language impairments. In addition, blockade of the striatal dopamine receptor leads to extrapyramidal side effects, causing tremors, muscle rigidity, and tics that interfere with the joint movements required for speech.

Therefore, voice and language are very good candidates as biomarkers in monitoring both symptoms and treatment effects in schizophrenia to detect onsets of relapses.

The aim of this study is to determine whether voice biomarkers can be used to objectively monitor symptoms and treatment effects in schizophrenia in order to detect onset of relapses.

ELIGIBILITY:
Inclusion Criteria:

* Affiliated to a social security or other social protection scheme
* Diagnosed with schizophrenia according to the DSM-5 (code F20)
* Stable state without duration criteria
* Main treatment with risperidone or paliperidone, aripiprazole, olanzapine in oral or long-acting injectable form
* Complementary treatment with an antipsychotic for anxiolytic or sedative purposes: chlorpromazine, loxapine or cyamemazine
* Able to speak and read French
* Able to perform speech evaluations
* Able to answer questionnaires on smartphone
* May be under curatorship or guardianship
* Agreeing to participate in the study and with informed consent signed by the subject, as well as by the legal representative in the case of a person under curatorship or guardianship

Exclusion Criteria:

* Suffering from a pathology that impairs French
* Suffering from a neurological pathology: multiple sclerosis, Parkinson's disease, Huntington's disease or neurodegenerative disease
* Treatment with lithium salts
* Anti-epileptic treatment
* Participant in another study involving medication

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2026-10-04 (Estimated); Study Completion 2026-10-04 (Estimated)

PRIMARY OUTCOMES:
Voice interviews recorded on Callyope application | Month 0, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6
  The analysis of the interviews (acoustic and linguistic features) will be implemented in a voice model predicting a score.
Plasma concentration of antipsychotics | Month 0, Month 2, Month 4, Month 6
  Plasma concentration of antipsychotics measured in ng/mL from Month 0 to Month 6.

SECONDARY OUTCOMES:
Age | Month 0
  Age in years
Weight | Month 0
  Weight in kilograms
Sex | Month 0
  Sex (Male / Female)
Change from Baseline in the schizophrenia severity | Month 0, Month 2, Month 4, Month 6
  Schizophrenia severity will be assessed by the investigator with PANSS (Positive and Negative Syndrome Scale) scale. For positive symptoms, score range is 7-49; For negative symptoms, the score range is 16 to 112. Higher score mean a worse outcome.
Change from Baseline in the schizophrenia severity | Month 0, Month 2, Month 4, Month 6
  Schizophrenia severity will be assessed by the investigator with CGI-SH (Clinical Global Impression - Schizophrenia) scale.
  Score range (min - max): 0 - 7 for the severity subscale Symptomatic remission correspond to a score ≤3 (CGI-S).
Changes from Baseline in the schizophrenia severity | Month 0, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6
  Schizophrenia severity will be assessed by the investigator with the scores from MCSI (Modified version of the Colorado Symptom Index) questionnaire.
  Score range (min-max) : 5-70 Higher score relates to worse outcome
Number of hospitalizations | From enrollment to the end of study at 6 months
  The total number of schizophrenia-related hospitalizations will be collected by the investigator from enrollment to the end of study at 6 months.
Total sleep duration | From enrollment to the end of study at 6 months
  The total sleep duration in hours and minutes will be automatically measured by the Callyope application
Duration of daily physical activity | From enrollment to the end of study at 6 months
  Duration of time spent at home, time in stationary mode in hours and minutes automatically assessed by the Callyope application
Phases of sleep duration | From enrollment to the end of study at 6 months
  Duration of sleep phases in hours and minutes automatically assessed by the Callyope application
Plasma concentration of sedative antipsychotics | Month 0, Month 2, Month 4, Month 6
  Plasma concentration of sedative antipsychotics measured in ng/mL from Month 0 to Month 6
Daily travel distance | From enrollment to the end of study at 6 months
  Maximum daily travel distance from home in kilometers automatically assessed by the Callyope application
Changes from Baseline in the symptoms (Depression, anxiety, functional autonomy, fatigue) | Month 0, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6
  Symptoms will be assessed by the score of the PHQ-9 (Patient Health Questionnaire - 9) questionnaire.
  Score range (min - max): 0 - 27 Higher score relates to a worse outcome
Changes from Baseline in feelings of loneliness or social isolation | Month 0, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6
  Feelings of loneliness or social isolation will be assessed by the investigator from the Score from UCLA 3-item Loneliness Scale.
  The total score ranges from 20 to 80. Higher scores indicate higher loneliness.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre De Maricourt, Dr, Principal Investigator — GHU Paris Psychiatry & Neurosciences
Locations (2):
- France (2):
  - Groupe Hospitalo-Universitaire Paris Psychiatrie et Neurosciences, Paris, Paris, Paris
  - Groupe Hospitalo-Universitaire Paris Psychiatrie & Neurosciences, Paris

IPD SHARING:
Plan to Share IPD: No